CLINICAL TRIAL: NCT02666404
Title: Impact of Amount of Fluid for Circulatory Resuscitation on Renal Function in Patients in Shock: Evaluating the Combination of Intraabdominal Pressure and Renal Resistive Index With Hemodynamic Parameters for Guidance of Shock Therapy - A Multicenter International Clinical Trial
Brief Title: Impact of Amount of Fluid for Circulatory Resuscitation on Renal Function in Patients in Shock
Acronym: VoluKid
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Volume resuscitation procotol has changed around 2017/2018 to less volume/more vasopressors.
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EKNZ 2015-401
Record Dates: First submitted 2016-01-18; First posted 2016-01-28 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Shock
Keywords: Volume Resuscitation; Shock; Body Impedance Measurement; Renal Resistive Index; Acute Kidney Injury; Renal Replacement Therapy
MeSH Terms: conditions — Shock; Acute Kidney Injury | interventions — Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Volume Resuscitation (Experimental): We would like to establish new endpoints for guidance of volume resuscitation by implementing new measurements (body impedance, renal resistive index).
  Interventions: Other: Measurement

INTERVENTIONS:
Other: Measurement — We will perform those new measurements and assessments for guidance of fluid resuscitation at 0, 6, 24, 48, and 72 hours after shock diagnosis and concomitant fulfillment of eligibility requirements
  Other Names: Body Impedance Measurement; Renal Resistive Index; Intra-abdominal Pressure

SUMMARY:
Volume resuscitation is the mainstay of treatment in most types of shock, especially in hemorrhagic and septic shock. Septic shock is a main cause of morbidity and mortality worldwide. Although there has been a lot of research to evaluate optimal amount and composition of fluids for volume resuscitation (e.g. colloids, crystalloids, red blood cell transfusion, albumin, fresh frozen plasma) particularly in the past decade, results remain inconclusive and to some extent contradictive. The investigators would like to contribute to the establishment of new endpoints for the guidance of shock therapy focusing on the first 24 and 48 hours, amending the currently used parameters (i.e. cardiac output, heart rate, blood pressure, central venous pressure) with new measurements (see study specific measurements). The goal is to decrease the need for renal replacement therapy, thereby eventually reducing patient morbidity and mortality.

DETAILED DESCRIPTION:
Background and Rationale, clinical evidence to date:

All forms of shock and especially septic shock, in which tissue metabolic demands are not fulfilled by blood supply, are main causes of morbidity and mortality worldwide and develops in one third of the patients admitted to the ICU. Not only is this high incidence alarming, the uncertainty about the undeceiving parameters for guidance of fluid resuscitation to not only avoid acute kidney injury and renal replacement therapy but also the consequences of fluid overload, such as interstitial pulmonary edema, underline the importance of further research within this field. This is why the investigators would like to contribute to the establishment of new parameters for the guidance of shock therapy focusing on the first 72 hours, amending the currently used parameters (i.e. cardiac output, heart rate, blood pressure, central venous pressure) with new measurements, including assessment of total body water, renal vascular resistance (renal resistive index (RRI)) and microcirculatory blood flow.

Although the application of intravenous crystalloid fluids, red blood cell concentrates in anemia, and catecholamines or inotropes are the mainstay of shock therapy, no clear endpoints for the fluid resuscitation or the hemodynamic endpoints for catecholamine therapy have been established so far. Static parameters such as central venous or arterial pressure, cardiac output, or plasma lactate failed in the guidance of the amount of fluid administered. The administration of intravenous fluids in response to so-called dynamic tests, such as stroke volume variation in response to fluid bolus administration, also did not show an influence on organ dysfunction and mortality due to shock. Acute kidney injury (AKI) is the most frequent organ dysfunction in patients in shock. Despite a more aggressive early fluid resuscitation and correction of arterial blood pressure, the incidence of AKI does not seem to decrease. One possible reason is that the excessive amount of fluid administered to these patients for hemodynamic stabilization and maintenance of urinary output harm kidney function. Indeed, a correlation between total amount of fluid administered, high central venous pressure, organ dysfunction, and mortality has been shown in patients with severe sepsis and septic shock. Established static and dynamic hemodynamic parameters are not influenced by the severity of capillary leakage and microcirculatory impairment due to inflammation-induced injury in capillaries. The relatively low perfusion pressure together with interstitial edema, microcirculatory injury, and a high outflow pressure may harm renal function by a decreased glomerular urine excretion. Intraabdominal pressure, total body water, and central venous pressure together with the renal resistive index may be additional measurements to reduce the rate of acute kidney injury and to guide fluid therapy in shock.

The goal of the present study is to refine fluid resuscitation endpoints with new measurements to administer the optimal amount of fluid with the smallest possible adverse effects. Complexity of therapy in severe sepsis and septic shock as well as in other shock states was the topic of numerous studies showing no benefit of advanced macro-circulatory parameters for guidance of fluid resuscitation in shock. If the chosen measurements are unable to establish new endpoints for guidance in shock therapy, the investigators' research might be expanded to the evaluation of future therapies, such as biomarkers or stem cells. After establishment of more regional resuscitation endpoints, the investigators plan to evaluate these endpoints in a randomized, controlled setting against established hemodynamically-guided shock therapy.

Investigational measurements:

The investigators will perform the following new measurements and assessments for guidance of fluid resuscitation at 0, 6, 24, 48, and 72 hours after shock diagnosis and concomitant fulfillment of eligibility requirements:

Patient characteristics:

* Sepsis-related Organ Failure Assessment (SOFA) score, daily
* APACHE II score, first 24 hours
* Simplified Acute Physiology (SAPS) II score, first 24 hours

Established parameters:

* Hemodynamic parameters (cardiac index [5], central venous pressure, blood pressure, heart rate, central/mixed venous oxygen saturation = ScvO2/venous oxygen saturation (SvO2), pulmonary capillary occlusion pressure (PAOP)
* Use of inotropic and vasoactive drugs (epinephrine, norepinephrine, milrinone, dobutamine, levosimendan)
* Laboratory parameters (lactate, sodium, potassium, blood sugar concentration and need for insulin therapy with respect to need for immunosuppressive therapy)
* Parameters of renal function (creatinine, creatinine clearance, blood urea nitrogen, urine output, potassium, urinary protein, urinary sediment analysis, sodium excretion fraction, need for renal replacement therapy)

  * Creatinine clearance after 24, 48, and 72 hours
  * Urinary sediment analysis 72 hours
  * Urinary protein screening after 72 hours

Fluid administration:

* Total amount of fluids (ml) administered
* Total amount of crystalloids (ml) administered after onset of shock symptoms
* Total amount of colloids (ml) administered
* Amount of red blood cell and plasma transfusion
* Amount of albumin infusion

Alternative parameters influenced by severity of capillary leakage and microcirculatory injury:

* Renal artery resistive index (Doppler analysis)
* Intra-abdominal pressure (bladder pressure management)
* Total body water (bio-impedance analysis): this is a commonly used method for assessment of body composition
* Microcirculatory blood flow (CytoCam incident dark-field illumination): "hand-held device (…), providing new means of directly visualizing the microcirculation and evaluating the effects of interventions on microcirculatory flow in easily accessible surfaces"

Outcome parameters:

* Acute kidney injury according to 'Kidney Disease: Improving Global Outcomes' (KDIGO) criteria
* Need for renal replacement therapy
* Length of intensive care stay
* Length of hospital stay

Safety: risks and benefits:

Since the investigators are only performing noninvasive measurements, additional to interventions, pharmacotherapy and measurements in shock patients, there will be no contributing risk by study enrolment. Since there will be a more precise way for guidance of fluid resuscitation in shock evoked by these study-specific measurements (bio-impedance analysis, doppler analysis, CytoCam incident darkfield illumination), study patients might even benefit from enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* State of shock (any type) upon admittance to the ICU.

Exclusion Criteria:

* Age below 18 years
* Non-shock state
* Terminal state
* Pregnancy
* Jehovah's Witnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury (KDIGO staging for severity of acute kidney injury ). | Assessment at 0, 6, 24, 48, and 72 hours after shock diagnosis
  Change in renal function from baseline according to KDIGO staging

SECONDARY OUTCOMES:
Difference in lactate values (µmol/l) | Between 6 and 24 hours after admittance to the ICU and baseline (t1/t2 - t0)
Need for renal replacement therapy (KDIGO staging for severity of acute kidney injury) | Assessment at 0, 6, 24, 48, and 72 hours after shock diagnosis
Length of ICU stay | 1 month
  If Patient stay exceeds one month, we will assess the data at intervals of one month
Length of hospital stay | 1 month
  If Patient stay exceeds one month, we will assess the data at intervals of one month
Need for mechanical ventilation | During 27 hours
In-hospital, 30-, and 90-day mortality | 0-90 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin Siegemund, MD, Study Chair — Deputy Chief Physician, Surgical Intensive Care Unit
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Average Acute Physiology And Chronic Health Evaluation (APACH) II score/SAPS II score/SOFA score/KDIGO criteria